CLINICAL TRIAL: NCT05556460
Title: A Prospective, Multicenter, Parallel, Randomized Controlled Study to Evaluate the Safety and Effectiveness of the DragonFly-T Transcatheter Tricuspid Valve Clip System in the Treatment of Tricuspid Regurgitation
Brief Title: Safety and Effectiveness Study of DragonFly-T System for Severe Tricuspid Regurgitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Valgen Medtech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF-VL-03
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency | interventions — Nutrition Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomized - Device Group (Experimental): The experimental group is allocated to use a novel tricuspid valve repair system for edge-to-edge repair manufactured by Hangzhou Valgen Medtech Co., Ltd. and will continue to be managed on medical therapy, per physician discretion
  Interventions: Device: DragonFly-T Transcatheter Tricuspid Valve Repair System
- Randomized - Control Group (Active Comparator): Subjects will continue to be managed on medical therapy, per physician discretion
  Interventions: Drug: Medical therapy

INTERVENTIONS:
Device: DragonFly-T Transcatheter Tricuspid Valve Repair System — To conduct edge-to-edge repair with DragonFly-T System under the guidance of transesophageal echocardiography.
  Arms: Randomized - Device Group
Drug: Medical therapy — Subjects will continue to be managed on medical therapy, per physician discretion
  Arms: Randomized - Control Group

SUMMARY:
The primary objective of this trial is to demonstrate the safety and effectiveness of the DragonFly-T system in improving clinical outcomes in symptomatic patients with severe tricuspid regurgitation (TR), who are at intermediate or greater estimated risk for mortality or morbidity with tricuspid valve surgery. This randomized controlled trial will compare the investigational device (DragonFly-T system) to Control (Medical Therapy).

DETAILED DESCRIPTION:
A Prospective, Multicenter, Parallel, Randomized Controlled Study to Evaluate the Safety and Efficacy of the DragonFly-T Transcatheter Tricuspid Valve Clip System in the Treatment of Tricuspid Regurgitation. After signing the informed consent form, participants in the experimental group will be treated with the Dejin Medical DragonFly-T Transcatheter Tricuspid Valve Clip System and continue receiving medical therapy as determined by the investigator. Participants in the control group will continue to receive medical therapy as determined by the investigator. Control group participants are allowed to cross over to the experimental group after completing the 12-month follow-up. All participants will undergo clinical follow-up before discharge (not applicable to control group participants), at 30 days post-treatment, 6 months post-treatment, 12 months post-treatment, and annually at 2, 3, 4, and 5 years..

The primary endpoint is the hierarchical composite endpoint formed by all-cause mortality or tricuspid valve reintervention, heart failure hospitalization, and KCCQ improvement at 12 months post-treatment.

To evaluate the safety and effectiveness of the Valgen Medtech DragonFly-T Transcatheter Tricuspid Valve Repair System in the treatment of patients with severe tricuspid regurgitation (TR), who are at intermediate or greater estimated risk for mortality or morbidity with tricuspid valve surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. In the judgment of the local cardiac team, the patient has been adequately treated according to applicable standards (including medical management)and has been stable for at least 30 days.
3. Despite the drug optimization treatment according to the above method, patients still have symptoms of TR;
4. Determined by the local cardiac team to be at intermediate or higher risk for tricuspid valve surgery
5. New York Heart Association (NYHA) Cardiac function Class II-IVa;

5. The patient is suitable for transcatheter tricuspid valve repair, suitable for the use of this study instrument, and the femoral vein access is feasible and can accommodate catheter; 6. Patient must provide written informed consent before any steps related to the study.

Exclusion Criteria:

1. Tricuspid valve leaflet anatomy, which may preclude clip implantation, proper clip positioning on the leaflets, including but not limited to the following:

   1. Evidence of calcification in the grasping area;
   2. Presence of a severe coaptation defect of the tricuspid leaflets;
   3. Severe leaflet defect(s) and cleft preventing proper device placement determined by ECL;
   4. Epstein anomaly.
2. Other serious heart valvular diseases requiring intervention or planning to intervention in the next 12 months; Note: If mitral and tricuspid valve lesions are combined, mitral valve surgery can be performed first, and re-evaluation can be performed 60 days after surgery.
3. Tricuspid stenosis evaluated by ECL and/or cross-tricuspid differential pressure ≥ 5 mmHg;
4. Previous tricuspid valve surgery or transcatheter therapy;
5. Echocardiography suggested intracardiac thrombus, tumor or mass, or femoral vein and inferior vena cava implants or thrombus;
6. TTE and TEE are unable to evaluate tricuspid valve anatomy; Participated in any drug and/or medical device clinical trials within 1 month prior to the trial; ……

28. The researchers do not consider it appropriate to be enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2027-08-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Hierarchical Composite of All-cause Death or Tricuspid Valve Intervention, Heart Failure Hospitalizations, and KCCQ Improvement | 12 months

SECONDARY OUTCOMES:
Tricuspid regurgitation severity | 30 days, 6 months, and 12 months
  Percentage of patients with tricuspid regurgitation of 2+ or less.
Change in 6 minutes walk test distance | 30 days, 6 months, and 12 months
  Improvement in 6 Minute Walk Test distance
Quality of life improvement | 30 days, 6 months, and 12 months
  Improvement in quality of life (QoL) , as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ).
Acute procedural success | Immediately after procedure, Discharge: The day after the patient's exit from the cardiac catheterization laboratory
Acute device success | Immediately after procedure
Incidence of major adverse events (MAEs) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jian'an Wang, MD, PH.D, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (2):
- China (2):
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No